CLINICAL TRIAL: NCT07276490
Title: The Pacing in Atrioventricular Block: a Comparative Evaluation of Central Haemodynamics, Cardiac Function, and Quality of Life
Brief Title: Central Haemodynamics and Pacing for AV Block
Acronym: PACE-CCQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Collaborators: North Estonia Medical Centre (Other); Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Silver Heinsar, Clinical researcher, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 405/M-27
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Atrioventricular Block; Pacing Therapy; Right Ventricular Pacing; Conduction System Pacing
Keywords: conduction system pacing; atrioventricular block; right ventricular pacing
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right ventricular pacing (Active Comparator)
  Interventions: Device: Right ventricular pacing
- Conduction system pacing (Experimental)
  Interventions: Device: Conduction system pacing

INTERVENTIONS:
Device: Right ventricular pacing — Pacemaker implantation with RV lead placement
  Arms: Right ventricular pacing
Device: Conduction system pacing — Pacemaker implantation with conduction system (LBBAP) lead placement
  Arms: Conduction system pacing

SUMMARY:
A randomized, single-blind study comparing two pacing strategies in patients with atrioventricular block requiring permanent pacemaker implantation. This trial evaluates the impact of conduction system pacing (left bundle branch area pacing) versus standard right ventricular pacing on central hemodynamics, cardiac function, and patient quality of life over 12 months. The study will enroll 124 patients from two Estonian tertiary hospitals and measure central systolic arterial pressure as the primary outcome, with secondary assessments of arterial stiffness, echocardiographic parameters, electrical activation patterns, and quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Diagnosis of atrioventricular block
* Expected survival >1 year

Exclusion Criteria:

* Reduced left ventricular ejection fraction (EF <45%)
* Expected ventricular pacing burden <20%
* Inter-arm systolic blood pressure difference >15 mmHg
* Percutaneous coronary intervention or coronary artery bypass surgery within the last 30 days
* Secondary hypertension
* Orthostatic hypotension
* Clinically significant valvular heart disease
* Congenital heart disease
* Pulse wave analysis or pulse wave velocity measurement cannot be reliably performed
* Pregnancy or breastfeeding
* Withdrawal of consent by the subject
* Loss of contact during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Central systolic blood pressure | One year post implantation of pacemaker

CONTACTS AND LOCATIONS:
Locations (1):
- North Estonia Medical Centre, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: No